CLINICAL TRIAL: NCT03689296
Title: Patient-caregiver Collaboration for Better Cardiovascular Care for Patients With Long-term Mental Disorders: Multicentre Qualitative and Feasibility Studies
Acronym: COPsyCAT
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: DENIS PREPS 2017
Record Dates: First submitted 2018-09-17; First posted 2018-09-28 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Long-term Mental Disorders
MeSH Terms: interventions — Surveys and Questionnaires; Clinical Trials, Phase III as Topic; Focus Groups; Clinical Trials, Phase II as Topic; Clinical Trials, Phase I as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Users: Person with a long-term mental disorder
  Interventions: Other: Questionnaires (Phase 3); Other: Focus groups (Phase 2); Other: semi-structured interviews (Phase 1)
- Caregivers: Adult helping a person with a long-term psychological disorder
  Interventions: Other: Focus groups (Phase 2); Other: semi-structured interviews (Phase 1)
- Primary care professionals: Primary care professional in practice following at least one person with a long-term mental disorder
  Interventions: Other: Focus groups (Phase 2); Other: semi-structured interviews (Phase 1)
- Psychiatric professionals: Psychiatric specialist working in a hospital or in private practice
  Interventions: Other: Focus groups (Phase 2); Other: semi-structured interviews (Phase 1)

INTERVENTIONS:
Other: Questionnaires (Phase 3) — * CardioVascular Risk (CVR) questionnaire representation
  * SF12
  * Getting Better My Way
  * My recovery plan
  * Psycom
  * Partner In Health scale
  Groups: Users
Other: Focus groups (Phase 2) — Focus group interviews conducted by two health sociologists in 4 distinct categories: caregivers, patients, primary health care professionals and psychiatric professionals.
Other: semi-structured interviews (Phase 1) — Conduct of exploratory semi-directive interviews with users, caregivers, primary health care professionals and psychiatric professionals by a health sociologist

SUMMARY:
People with severe and persistent mental disorders (or SMI, Severe Mental Illness) have a life expectancy which is 20 years less than the general population, mainly due to excess mortality related to cardiovascular disease. Moreover, despite an overall increase in life expectancy, the gap is widening between people with long-term psychological disorders and the general population.

This early excess mortality is explained by disparities between people with SMI and the general population not only in access to and use of health services but also in the quality and type of care provided. There is also an over-representation of risk factors and cardiovascular pathologies regardless of the mental disorder, despite the current recommendations for best practices.

The World Health Organization has defined the fight against somatic comorbidities as one of the axes of the European Mental Health Plan and one of the reference themes of the World Health Organization Mental Health Evidence and Research Programme (EPSM-Lille-Métropole). The Groupement de Coopération Sanitaire pour la recherche et la formation en santé mentale, which brings together 17 hospitals in France and relays the actions of the World Health Organization's Collaborating Centre, has decided to make it into a national research project.

Moreover, it is recognized that "medical" management of a disease is all the more effective when the patient is involved. However, the empowerment of people with long-term psychological disorders has never been put at the centre of a strategy to reduce cardiovascular risk.

In this context, we hypothesize that one of the keys to reducing cardiovascular risk would be to take into account the experience and representations of this risk by all stakeholders (people with long-term psychological disorders, their carers, primary health professionals and psychiatric professionals).

ELIGIBILITY:
Inclusion Criteria:

1. For all groups:

   * Adult person,
   * Person who has given his or her consent to participate in the study, with the consent of the tutor in the context of guardianship,
   * Fluent use of the French language,
2. For the "Users" group:

   - Person with a long-term psychological disorder: Long-term illness (ALD 23), followed by outpatient or full hospitalization
3. For the "Caregivers" group:

   - Adult helping a person with a long-term psychological disorder with a Long-Term Disability (ALD 23) and who has given his or her consent to be contacted for the study,
4. For the "Primary Care Professionals" group:

   - Primary care professional in practice following at least one person with a long-term psychological disorder with a Long-Term Disability (ALD 23),
5. For the "Psychiatric Professionals" group - Professional currently in practice who is part of a psychiatry team or in private practice

Exclusion Criteria:

1. For all groups:

* Person who is physically or psychologically unable to participate in the focus group and/or program at the time of the study
* Person not affiliated to the National Health Insurance
* Objection to participation by the patient or his legal representative, carers and health professionals.
* Patient under guardianship
* Patient who participated in Phase 1 or 2 of the study
* Patient not able to attend the 6-month visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients followed in ambulatory or full hospitalization (depending study phase)
Sampling Method: Non-Probability Sample
Enrollment: 127 (Actual)
Dates: Start 2019-06-27 (Actual); Primary Completion 2024-08-07 (Actual); Study Completion 2024-08-07 (Actual)

PRIMARY OUTCOMES:
Focus group interview completion | Through study completion, an average of 14 months

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourogne, Dijon, France

REFERENCES:
- [Derived] Baleige A, Besnard JF, Meunier-Beillard N, Demassiet V, Monnier A, Ouezini A, Lambert O, Charrel C, Mazas O, Oberlin J, Roelandt JL, Denis F. A collaboration between service users and professionals for the development and evaluation of a new program for cardiovascular risk management in persons with a diagnosis of severe mental illness: French multicenter qualitative and feasibility studies. Int J Ment Health Syst. 2019 Dec 27;13:74. doi: 10.1186/s13033-019-0331-6. eCollection 2019. PMID 31889999